CLINICAL TRIAL: NCT05320406
Title: Mechanism and Predictors of Cardiotoxicity After Prostate Cancer Treatment: A Parallel Cohort and Randomized Trial Comparing Radiation Alone, Radiation Plus Leuprolide, and Radiation Plus Relugolix
Brief Title: RElugolix VErsus LeUprolide Cardiac Trial
Acronym: REVELUTION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Prostate Cancer Foundation (Other)
Responsible Party: Principal Investigator, Sagar Patel, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003654; NCI-2022-00117 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00003654; RAD5484-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); 22YOUN21 (Other Grant/Funding Number: Prostate Cancer foundation)
Record Dates: First submitted 2022-03-18; First posted 2022-04-11 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Localized Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated; Proton Therapy; Brachytherapy; Radiosurgery; Leuprolide; relugolix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm I (radiation therapy alone) (Active Comparator): Patients undergo definitive radiation therapy alone (IMRT, SBRT, proton therapy, brachytherapy) in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation therapy
- Arm II (radiation therapy plus leuprolide) (Experimental): Patients undergo radiation therapy as in Arm I and receive leuprolide SC or IM every 3 or 6 months. Treatment continues for 6 to 12 months (depending on risk) in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation therapy; Drug: Leuprolide
- Arm III (radiation therapy plus relugolix) (Experimental): Patients undergo radiation therapy as in Arm I and receive relugolix PO QD. Treatment continues for 6 to 12 months (depending on risk) in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation therapy; Drug: Relugolix

INTERVENTIONS:
Radiation: Radiation therapy — Undergo radiation therapy
  Other Names: External beam radiation therapy; Intensity modulated radiation therapy; Proton therapy; Brachytherapy; Stereotactic body radiotherapy
Drug: Leuprolide — Given IM or SC
  Other Names: Leuprolide acetate; Lupron
  Arms: Arm II (radiation therapy plus leuprolide)
Drug: Relugolix — Given PO
  Other Names: Orgovyx; TAK-385
  Arms: Arm III (radiation therapy plus relugolix)

SUMMARY:
This clinical trial investigates the impact of prostate cancer treatment, specifically androgen deprivation therapy (ADT), on the heart and coronary vessels among men with localized, non-metastatic prostate cancer undergoing definitive radiation therapy and concomitant ADT. Recently, cardiovascular toxicity from hormone therapy that is routinely used for prostate cancer (e.g. leuprolide) has emerged as a concern, yet studies identifying who is at risk and the mechanism of cardiac damage are lacking. Additionally, a new hormone therapy drug, relugolix, has recently been Food and Drug Administration (FDA)-approved and may reduce toxicity to the heart. This trial intends to investigate the mechanism of cardiovascular toxicity from ADT, investigate the mechanism by which relugolix reduces cardiovascular toxicity, and identify predictive biomarkers to improve individualized risk-assessment for cardiovascular toxicity from ADT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify and compare the association of gonadotrophin releasing hormone (GNRH)-agonist leuprolide versus GNRH-antagonist relugolix with coronary atherosclerosis and progression in men with prostate cancer.

II. Determine the relationship between leuprolide versus relugolix with downstream immune effector response that is implicated in atherosclerosis.

II. Determine how pre-existing genomic alterations associated with proinflammatory immunity impact development of CV toxicity following GNRH-agonist (GNRHa) versus relugolix.

III. Identify imaging biomarkers associated with increased risk of CV toxicity from ADT

OUTLINE: Patients undergoing radiation therapy alone as part of their standard treatment are assigned to Arm I. Patients undergoing radiation therapy and ADT as part of their standard treatment are randomized to Arm II or Arm III.

ARM I: Patients undergo definitive radiation therapy in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo radiation therapy as in Arm I and receive leuprolide subcutaneously (SC) or intramuscularly (IM) every 3 or 6 months. Treatment continues for 6 to 24 months (depending on cancer risk) in the absence of disease progression or unacceptable toxicity.

ARM III: Patients undergo radiation therapy as in Arm I and receive relugolix orally (PO) once daily (QD) for 6 to 24 months (depending on risk) in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Men >= 18 years old
* Non-metastatic prostate cancer
* Non-metastatic, biochemically recurrent prostate cancer
* Plan to undergo curative-intent pelvic radiation therapy with or without ADT

Exclusion Criteria:

* Metastatic prostate cancer requiring > 24 months of ADT
* Prior exposure to androgen deprivation therapy
* Prior exposure to chemotherapy or immunotherapy
* History of cardiac bypass surgery or percutaneous coronary intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2026-10-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar A Patel, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (4):
- United States (4):
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Started | 29 | 34 | 31
Completed | 28 | 28 | 29
Not Completed | 1 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix) | Total
Number analyzed (Participants) | 29 | 34 | 31 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 7 | 27
  >=65 years | 19 | 24 | 24 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.79 (6.75) | 68.85 (8.12) | 68.81 (8.83) | 67.89 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 29 | 34 | 31 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 11 | 7 | 24
  White | 22 | 19 | 21 | 62
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 29 | 34 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: Total Coronary Plaque Volume in Major Coronary Arteries (i.e. Left Anterior Descending, Left Circumflex, Right Major Coronary Arteries)
Description: Using cardiac computed tomography angiography (CCTA), total coronary plaque volume will be determined using an artificial intelligence-enabled quantitative coronary plaque analysis (AI-QCPA) through a commercially available and validated software service (HeartFlow, Inc). Each coronary artery (right coronary, left main, left anterior descending, and left circumflex) will be scored, and plaque volumes were summed over all segments.
Time Frame: From baseline to 12 months post-treatment initiation
Measure: Median (95% Confidence Interval); unit: mm3
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Number analyzed (Participants) | 28 | 31 | 31
mm3
  Baseline | 103.0 [79.0 to 182.0] | 204.0 [73.0 to 556.5] | 272.0 [65.0 to 766.0]
  Month 12 | 130.0 [55.0 to 265.0] | 290.0 [153.0 to 655.5] | 265.0 [100.0 to 807.0]

2. Secondary Outcome: Non-calcified Coronary Plaque Volume in Major Coronary Arteries (i.e. Left Anterior Descending, Left Circumflex, Right Major Coronary Arteries)
Description: as for outcome 1
Time Frame: From baseline to 12 months post-treatment initiation
Measure: Median (95% Confidence Interval); unit: mm3
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Number analyzed (Participants) | 28 | 31 | 31
mm3
  Baseline | 98.0 [74.0 to 167.0] | 157.0 [65.5 to 464.5] | 206.0 [56.0 to 620.0]
  Month 12 | 112.0 [42.0 to 215.0] | 252.0 [133.0 to 511.0] | 236.0 [92.0 to 613.0]

3. Other Pre Specified Outcome: Calcified and Low-attenuation Coronary Plaque Volume in Major Coronary Arteries (i.e. Left Anterior Descending, Left Circumflex, Right Major Coronary Arteries)
Description: as for outcome 1
Time Frame: From baseline to 12 months post-treatment initiation
Measure: Median (95% Confidence Interval); unit: mm3
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Number analyzed (Participants) | 28 | 31 | 31
mm3
  Baseline | 11.5 [2.3 to 25.8] | 34.0 [5.8 to 98.8] | 41.0 [9.0 to 175.0]
  Month 12 | 13.0 [4.0 to 38.8] | 44.0 [12.3 to 109.0] | 46.0 [16.0 to 185.0]

4. Other Pre Specified Outcome: Coronary Artery Calcium Score (CACS)
Description: The CACS will be measured by the Agatston score (range 0-400, with higher scores indicating more coronary artery calcium) on precontrast cardiac computed tomography anigiography (CCTA) scans by two blinded, board-certified cardiologists.
Time Frame: From baseline to 12 months post-treatment initiation
Measure: Median (95% Confidence Interval); unit: Agatston score (range 0-400)
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Number analyzed (Participants) | 28 | 31 | 31
Agatston score (range 0-400)
  Baseline | 24.9 [5.3 to 91.3] | 106.6 [4.5 to 249.6] | 96.0 [14.0 to 390.1]
  Month 12 | 36.0 [6.8 to 101.8] | 102.7 [19.9 to 262.5] | 109.8 [31.8 to 509.3]

5. Other Pre Specified Outcome: Number of Participants With <30%, 30-49%, 50-69%, and >70% Maximum Coronary Vessel Stenosis at Baseline and Month 12
Description: Coronary computed tomographic angiography post-contrast images were used for vessel stenosis, using an artificial intelligence-informed coronary stenosis quantification tool (AI-CSQ, Roadmap Analysis, Heart flow, Mountain View CA). Stenoses regions are defined in ranges of 0-29%, 30-49%, 50-69%, and >70%. The number of participants within each treatment meeting these stenosis thresholds were quantified at baseline and month 12.
Time Frame: From baseline to 12 months post-treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Number analyzed (Participants) | 28 | 31 | 31
Participants
  Baseline: <30% | 5 | 3 | 4
  Baseline: 30% - 49% | 12 | 9 | 8
  Baseline: 50% - 69% | 9 | 15 | 16
  Baseline: 70% - 99% | 2 | 4 | 3
  Month 12: <30% | 6 | 2 | 6
  Month 12: 30% - 49% | 10 | 8 | 6
  Month 12: 50% - 69% | 10 | 17 | 15
  Month 12: 70% - 99% | 2 | 4 | 4

6. Other Pre Specified Outcome: Major Adverse Cardiovascular Events
Description: Incidence of myocardial infarction, need for coronary revascularization, and/or sudden cardiac death will be measured for up to 2 years following enrollment.
Time Frame: From baseline to at least 2 years post-treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Number analyzed (Participants) | 28 | 31 | 31
Participants | 1 | 3 | 0

7. Other Pre Specified Outcome: Testosterone Kinetics
Description: Change in total testosterone levels (ng/dL) will be measured at baseline and month 0, 3, 6, and 12 between treatment arms. Testosterone change over time will be summarized and plotted over time for each treatment arm.
Time Frame: Baseline and month 0, 3, 6, 12
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
Number analyzed (Participants) | 28 | 31 | 31
ng/mL
  0 | 254.433 (16.365) | 292.735 (15.114) | 254.548 (15.828)
  3 | 266.358 (16.633) | 37.483 (10.254) | 26.468 (7.325)
  6 | 260.606 (17.815) | 31.063 (8.018) | 25.538 (5.325)
  12 | 253.631 (18.149) | 142.007 (18.503) | 199.673 (16.573)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm I (Radiation Therapy Alone) | Arm II (Radiation Therapy Plus Leuprolide) | Arm III (Radiation Therapy Plus Relugolix)
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 23/28 | 27/31 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Radiation Therapy Alone) (N=28) | Arm II (Radiation Therapy Plus Leuprolide) (N=31) | Arm III (Radiation Therapy Plus Relugolix) (N=31)
sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Radiation Therapy Alone) (N=28) | Arm II (Radiation Therapy Plus Leuprolide) (N=31) | Arm III (Radiation Therapy Plus Relugolix) (N=31)
Cystitis noninfective (Renal and urinary disorders) | 6 (6) | 13 (16) | 12 (14)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 10 (14) | 14 (24)
Fatigue (General disorders) | 9 (13) | 22 (33) | 26 (29)
Hot flashes (Vascular disorders) | 0 (0) | 18 (27) | 20 (24)
Urinary frequency (Renal and urinary disorders) | 12 (14) | 22 (24) | 24 (29)
Urinary retention (Renal and urinary disorders) | 9 (11) | 14 (19) | 6 (6)
Urinary urgency (Renal and urinary disorders) | 10 (11) | 15 (19) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT05320406/Prot_SAP_002.pdf
  • Informed Consent Form (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT05320406/ICF_001.pdf